CLINICAL TRIAL: NCT03099057
Title: Study of Prognostic Factors in Interventional Rhythmology
Acronym: PRINT
Status: Terminated | Type: Observational
Why Stopped: Lake of personnel
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC16.0104
Record Dates: First submitted 2017-03-17; First posted 2017-04-04 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Cardiac Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: follow-up of patients after interventional rhythm operation — The follow-up will take place at 3 months postoperatively, then at 1 year and then annually for 5 years.

SUMMARY:
Develop a prospective register assessing the short- and long-term complications of patients undergoing interventional rhythm

DETAILED DESCRIPTION:
To assess the fate of patients who have undergone a technical procedure at the Cardiology Plate (implantation / extraction of a pacemaker, a defibrillator, radiofrequency ablation or cryo-ablation, left auricle closure, electro- Physiological exploration), and to determine prognostic factors / markers in this population.

ELIGIBILITY:
Inclusion Criteria:

Patient to undergo:

* Implantation of a cardiac pacemaker or cardiac defibrillator or
* Extraction of pacemaker / defibrillator housing or probes or
* Realization of a radiofrequency / cryo-ablation:
* Atrial fibrillation
* Focus of ventricular tachycardia
* An accessory or
* Any electrophysiological exploration or
* Installation of Holter implantable or
* Left auricular closure percutaneously Having formulated its non-opposition

Exclusion Criteria:

* Minor
* Patient's refusal
* Patients under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient that must undergo a gesture of interventional rythmology in the Department of Cardiology of the CHRU of Brest
Sampling Method: Probability Sample
Enrollment: 2805 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
The occurrence of adverse clinical events | 5 years
  The occurrence of the following adverse clinical events: infectious, rhythmic complications, hemodynamic, mortality any causes and cardiovascular post--interventional and in the length-course

SECONDARY OUTCOMES:
duration of intervention | Day 1
  The duration of the operation of interventional rhythmology will be measured
dose of X-radiation used | Day1
  the dose of X-radiation used shall be measured
volume of used contrast agent | Day1
  The volume of used contrast agent will be measured
duration of hospitalization | 3 months
  the duration of hospitalization will be measured
need for reoperation | 5 years
  the need for reoperation will be assessed
evolution of the ECG | 5 years
  The evolution of the ECG will be estimated
evolution of the echocardiographic parameters | 5 years
  the evolution of the echocardiographic parameters will be estimated

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Mansourati, Professor, Principal Investigator — University Hospital, Brest
Locations (1):
- CHRU Brest, Brest, France